CLINICAL TRIAL: NCT03066752
Title: Cognitive Dysfunction in MS: Using Altered Brain Oscillation to Link Molecular Mechanisms With Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, E. Ann Yeh, Associate Scientist, Research Institute, The Hospital for Sick Children
Other Study IDs: 1000054117
Record Dates: First submitted 2017-01-03; First posted 2017-02-28 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Pediatric Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 7 pediatric-onset multiple sclerosis
- 7 non-patient healthy volunteers

SUMMARY:
Up to 65% of patients with multiple sclerosis (MS) experience cognitive dysfunction. Diminution of mental capacity has a pervasive and profound impact on their quality of life. Subtle changes in white matter predict cognitive changes in these patients but how this disrupts brain function remains unclear. Development of effective therapeutics to restore normal cognition hinges on elucidating these functional changes. The investigators seek to uncover the patho-physiological basis for cognitive decline in MS. The investigators hypothesize that cognitive decline originates from disrupted gamma oscillations and that gamma oscillations are disrupted by molecular changes triggered by demyelination.

ELIGIBILITY:
Inclusion Criteria (*applicable to controls):

1. Must be between 6 and 17 years and 11 months of age*;
2. Have a diagnosis of MS according to the revised McDonald diagnostic criteria and/or International Pediatric MS Study Group criteria;
3. Has English language knowledge at the level needed to complete clinical questionnaires (4th grade level).*

Exclusion Criteria (*applicable to controls):

1. Neurological comorbidity.*;
2. Relapses or requires treatment with steroids within 30 days from enrollment;
3. Is pregnant at the time of enrollment.*;
4. Has any metal parts in their body (i.e. Cochlear (ear) implant, metal braces (dental fillings are o.k.).*;
5. Is younger than 6 years of age.*;
6. Is older than 18 years of age.*;
7. Has prior history of traumatic brain injury, neurological disorder, cerebral palsy, developmental delay or learning disability.*;
8. Requires sedation for brain scanning.*;
9. Is claustrophobic, as brain scanning requires children to enter a tunnel in the MRI machine.*

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Seven patients who have pediatric-onset multiple sclerosis and 7 healthy (non-patient) children are expected to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
Neuronal responses during simple and choice reaction time tasks | 60 minutes
  Video-based eye tracking in the MEG
MRI scans of the brain, including Diffusion Tensor Imagine (DTI) | 90 minutes
Neurocognitive Testing | 90 minutes
  Penn Computerized Neurocognitive Battery
Neurological Exam - Standard physical exam performed by the neurologist to determine the Expanded Disability Status Scale (EDSS) score. | 20 minutes
Clinical Interview | 10 minutes
  Series of questions about the participant's demographic and clinical information including, current and past health, family history, and medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No